CLINICAL TRIAL: NCT01572571
Title: Focused Multiorgan Ultrasound in the Emergency Evaluation of Undifferentiated Hypotension
Brief Title: Ultrasound in Undifferentiated Hypotension
Acronym: US-UHP
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Volpicelli, Principal Investigator, San Luigi Gonzaga Hospital
Other Study IDs: SLG-182/2011
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Hypotension
Keywords: Emergency ultrasound; Focused ultrasound; Point-of-care ultrasound; Undifferentiated hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background

* Symptomatic undifferentiated hypotension represents a negative prognostic factor and the strongest predictor of in-hospital mortality.
* Misdiagnosis may lead to delayed or incorrect treatment of some life-threatening conditions.

Aim

- The aim of the study is to evaluate the feasibility and accuracy of a new bedside ultrasound method that consists in the focused imaging of the thorax, abdomen and leg veins, in emergency.

Methods

* Hypotensive (<100 mm/Hg) patients presenting to our emergency department, complaining of at least one of the neurologic, respiratory and cutaneous signs and symptoms of inadequate tissue perfusion, are prospectively studied by ultrasound-focused assessment of the heart, lungs, inferior vena cava, peritoneum, aorta and leg deep veins.
* On the basis of physical examination and ultrasound results, the operator declares the diagnostic hypothesis without influencing the attending physician and the following diagnostic procedure (which includes ultrasound, when needed).
* The diagnostic hypothesis is compared with the final diagnosis, obtained after the hospital route and discussed by a panel of three blinded experts (one radiologist, one cardiologist and one emergency physician).
* The statistical agreement is calculated by the k of Cohen with p-value, confidence intervals and raw agreement (Ra).

ELIGIBILITY:
Inclusion Criteria:

* Arterial pressure <100 mm/Hg at presentation
* At least one of the following symptoms:
* Unresponsive
* Syncope
* Impaired mental status
* Respiratory distress
* Severe malaise and fatigue

Exclusion Criteria:

* Patients undergoing cardiopulmonary resuscitation
* Trauma patients
* Electrocardiographic and clinical diagnosis of STEMI or NSTEMI
* Clear cause of shock that needs immediate intervention (hemorrhage, gastrointestinal bleeding, drugs overdose)
* Late evolution of shock state in a patient already treated with known diagnostic tests

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with undifferentiated hypotension
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Correlation between the ultrasound primary diagnosis and the clinical final diagnosis | Clinical judgment on the final diagnosis as deduced from all the data obtained after hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Volpicelli, MD, Principal Investigator — San Luigi Gonzaga Hospital
Locations (1):
- San Luigi Gonzaga University Hospital, Department of Emergency Medicine, Orbassano, Torino, Italy

REFERENCES:
- [Background] Atkinson PR, McAuley DJ, Kendall RJ, Abeyakoon O, Reid CG, Connolly J, Lewis D. Abdominal and Cardiac Evaluation with Sonography in Shock (ACES): an approach by emergency physicians for the use of ultrasound in patients with undifferentiated hypotension. Emerg Med J. 2009 Feb;26(2):87-91. doi: 10.1136/emj.2007.056242. PMID 19164614
- [Background] Jones AE, Tayal VS, Sullivan DM, Kline JA. Randomized, controlled trial of immediate versus delayed goal-directed ultrasound to identify the cause of nontraumatic hypotension in emergency department patients. Crit Care Med. 2004 Aug;32(8):1703-8. doi: 10.1097/01.ccm.0000133017.34137.82. PMID 15286547
- [Background] Rose JS, Bair AE, Mandavia D, Kinser DJ. The UHP ultrasound protocol: a novel ultrasound approach to the empiric evaluation of the undifferentiated hypotensive patient. Am J Emerg Med. 2001 Jul;19(4):299-302. doi: 10.1053/ajem.2001.24481. PMID 11447518
- [Background] Copetti R, Copetti P, Reissig A. Clinical integrated ultrasound of the thorax including causes of shock in nontraumatic critically ill patients. A practical approach. Ultrasound Med Biol. 2012 Mar;38(3):349-59. doi: 10.1016/j.ultrasmedbio.2011.11.015. Epub 2012 Jan 21. PMID 22266231